CLINICAL TRIAL: NCT03014583
Title: Prospective, Randomized Study Comparing Conventional, Burst And High Frequency (HF) Spinal Cord Stimulation (SCS) in Refractory Failed Back Surgery Syndrome (FBSS) Patients After a 32-contact Surgical Lead Implantation
Brief Title: Study Comparing Conventional, Burst and High Frequency (HF) Spinal Cord Stimulation (SCS) in Refractory Failed Back Surgery Syndrome (FBSS) Patients After a 32-contact Surgical Lead Implantation
Acronym: MULTIWAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-A01145-46
Record Dates: First submitted 2016-12-13; First posted 2017-01-09 (Estimated); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- HF/TCS/BURST (Experimental): HF/TCS/BURST
  Interventions: Device: Precision Spectra™ system
- HF/BURST/TCS (Experimental): HF/BURST/TCS
  Interventions: Device: Precision Spectra™ system
- BURST/HF/TCS (Experimental): BURST/HF/TCS
  Interventions: Device: Precision Spectra™ system
- BURST/TCS/HF (Experimental): BURST/TCS/HF
  Interventions: Device: Precision Spectra™ system
- TCS/BURST/HF (Experimental): TCS/BURST/HF
  Interventions: Device: Precision Spectra™ system
- TCS/HF/BURST (Experimental): TCS/HF/BURST
  Interventions: Device: Precision Spectra™ system

INTERVENTIONS:
Device: Precision Spectra™ system — Neurostimulation procedures

SUMMARY:
Chronic Back and/or Leg Pain (CBLP) after spinal surgical procedures, a condition commonly labelled Failed Back Surgery Syndrome (FBSS), affects between 15% and 40% of patients after a spine surgery. Treatment of this chronic condition by further operation or medical management has a heavy financial impact on health care systems.

Many studies have demonstrated the efficacy and economic value of Spinal Cord Stimulation (SCS) for chronic neuropathic pain, and randomized controlled trials (RCTs) have shown SCS to be a clinically effective adjunct to medical management. SCS has the advantages of being reversible and less invasive than surgery and may cause fewer issues over time than long-term pharmacological treatments.

Despite variable levels of success in the literature, approximately 30-55% of the patients treated with traditional SCS for neuropathic pain disorders will not receive adequate long term pain relief. Therefore, technical SCS system refinements, as well as new techniques have emerged.

Two new stimulation waveforms based on traditional SCS technology have appeared to further optimize the outcome for specific painful conditions;

* Burst stimulation mode: which generates constant-current stimuli with 5 spikes at 500 Hz per burst and pulse width and interspike intervals of 1 ms.
* High-frequency stimulation (from 1 to 10 kHz) mode.

Several studies have demonstrated the potential interest of these 2 new waveforms to treat FBSS patients compared to traditional SCS.

The Precision Spectra™ system allows MultiWave Technology by offering a broad spectrum of waveform options (from Tonic Conventional Stimulation (TCS), BURST stimulation to High Frequency stimulation (HF)).

To date, literature data comparing these 3 stimulation patterns is lacking but it is suggested the pain relief in some of non-responsive patients can be "recaptured" by increasing the SCS frequency to 500 Hz by BURST stimulation or beyond by HF stimulation. It seems important to conduct RCT in crossover, thanks to the new Precision SCS Stimulator, to compare the effects of these 3 different SCS modalities in FBSS patients and to determine which concept is the most effective in terms of pain reduction and energy consumption.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or ≤ 80 years.
* Subject has FBSS and does not require further surgery. For the purposes of this study, FBSS is defined as persistent or recurrent low back and leg pain of at least 6 months duration following at least one decompression and/or fusion procedure.
* Subject has persistent low back and leg pain despite other treatment modalities (pharmacological, surgical, physical, or psychological therapies) that have been tried and did not prove satisfactory or are unsuitable or contraindicated for the subject.
* Average global pain is ≥ 50 mm as assessed by the baseline VAS.
* With significant back, with mean intensity on a back pain VAS ≥ 50 mm (mean daily VAS score calculated on 5 consecutive days).
* Meeting the criteria for spinal cord stimulation test according to HAS guidelines (multidisciplinary consultation, psychological assessment, etc.).
* Subject is a candidate for SCS.
* Absence of active psychosis or history of serious psychotic illness requiring hospitalisation.
* Understands and accepts the constraints of the study.
* Free subject, not under temporary or permanent guardianship and not subject to subordination.
* Patients covered by French national health insurance.
* Patients who have given their written consent to the study after having received clear information.

Exclusion Criteria:

* Age < 18 years or > 80 years
* Subject is or has been treated with SCS, subcutaneous or peripheral nerve stimulation, an intrathecal drug delivery system, requires back surgery at the location related to his/her original back pain complaint or experimental therapies.
* Cause of low back pain accessible to etiological "mechanical" surgical treatment (discogenic low back pain, vertebral instability, spinal deformity, etc.).
* Subject had most recent back surgery less than 6 months ago.
* Presenting a surgical, anaesthetic or psychiatric contraindication to implantation of a spinal cord stimulation system.
* Based on the opinion of the principal or sub-investigator, the subject is unable to operate the SCS equipment.
* Subject has a life expectancy of less than 24 months beyond study enrolment.
* Absence of signature of the informed consent form.
* Patients not covered by French national health insurance.
* Subjects requiring closer protection, i.e. minors, pregnant women, nursing mothers, subjects deprived of their freedom by a court or administrative decision, subjects admitted to a health or social welfare establishment, major subjects under legal protection, and finally patients in an emergency setting.
* Pregnant women, nursing mothers, women of childbearing potential not using effective contraception (hormonal/barrier: oral, parenteral, percutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total ovariectomy).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Global Pain VAS Visual Analogic Scale (VAS) | Month 3
  Global pain intensity from 0 to 10.

SECONDARY OUTCOMES:
Leg and back Pain Visual Analogic Scale (VAS) | Inclusion, Implantation, Month 0, Month 1, Month 2, Month 3, Month 6, Month 9, Month 15
  Leg and back pain intensity from 0 to 10.
Oswestry Disability Index (ODI) | Inclusion, Implantation, Month 0, Month 1, Month 2, Month 3, Month 6, Month 9, Month 15
  Self-administered questionnaire with 10 items. These items comprise assessments concerning pain intensity, degree of disability for personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling. The score is between 0 and 100% for which 0% is the best score.
EuroQol 5-Dimension 5 items (EQ-5D-5L) | Inclusion, Implantation, Month 0, Month 1, Month 2, Month 3, Month 6, Month 9, Month 15
  EQ-5D is a generic quality of life scale that is not specific for low back pain. The scale comprises 5 questions assessing mobility, self-care, usual activities, pain/discomfort and anxiety/depression. A global index with a maximum score of 1 is calculated from the responses to these 5 dimensions by means of nomograms. The maximum score of 1 indicates the best possible quality of life.
Paraesthesia perception Visual Analogic Scale (VAS) | Implantation, Month 0, Month 1, Month 2, Month 3, Month 6, Month 9, Month 15
  Paraesthesia perception scale intensity from 0 to 10.
Adverse Events and Serious Adverse Events Collection | from Inclusion to Month 15 (End Of Study)
  Any harmful event occurring in a person participating in a clinical trial, which is not necessarily related to the clinical trial or to the medical device used in this clinical trial
Hospital Anxiety and Depression Scale (HADS) | Inclusion, Implantation, Month 0, Month 1, Month 2, Month 3, Month 6, Month 9, Month 15
  The HADS scale investigates symptoms of anxiety and depression and their severity. Each answer corresponds to a number between 0 and 3. Adding these numbers together gives a total score per column (anxiety and depression). If the score of a column is greater than or equal to 11, this means that you are suffering from anxiety or depression.
Lead Performance and Lead Selectivity | Implantation, Month 0, Month 1, Month 2, Month 3, Month 6, Month 9, Month 15
  Lead performance: Overlapped surface ratios between paraesthesia coverage and painful area.
  Lead specificity: Overlapped surface ratios between paraesthesia coverage and non-painful area, unwanted to be covered.
Patient satisfaction via Patient Global Impression of Change (PGIC) | Month 0, Month 1, Month 2, Month 3, Month 6, Month 9, Month 15
  The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment. Although widely used in chronic pain clinical trials, PGIC's validity has not been formally assessed. PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital, Poitiers, France

REFERENCES:
- [Derived] Billot M, Naiditch N, Brandet C, Lorgeoux B, Baron S, Ounajim A, Roulaud M, Roy-Moreau A, de Montgazon G, Charrier E, Misbert L, Maillard B, Vendeuvre T, Rigoard P. Comparison of conventional, burst and high-frequency spinal cord stimulation on pain relief in refractory failed back surgery syndrome patients: study protocol for a prospective randomized double-blinded cross-over trial (MULTIWAVE study). Trials. 2020 Aug 3;21(1):696. doi: 10.1186/s13063-020-04587-6. PMID 32746899